CLINICAL TRIAL: NCT06856993
Title: Early Evaluation of Exosome Multiomics and Clinical Prognosis in Patients With Sudden Death
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hao Sun, MD, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: 2021-SR-320
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Sudden Cardiac Death; Exosome Multiomics; Clinical Prognosis
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: standardized medical care of cardiac arrest — The standardized medical care for cardiac arrest includes early cardiopulmonary resuscitation (CPR), defibrillation, advanced cardiac life support (ACLS), post-resuscitation care, and continuous monitoring of the patient's vital functions.

SUMMARY:
Acute coronary syndrome (ACS) is one of the main causes of death. Worldwide, tens of millions of patients are hospitalized for coronary heart disease and ACS every year. ACS may show acute myocardial infarction, unstable angina pectoris, and even induce early arrhythmia, leading to sudden death. Sudden cardiac death (SCD) has a strong correlation with ACS. Data from clinical and autopsy studies and death certificates show that 62-85% of patients with out of hospital SCD have a history of ACS, 10% have other cardiac structural abnormalities, and 5% have no cardiac structural abnormalities. An SCD surveillance study from Ireland concluded that most cases occurred in families, and the successful recovery of SCD was mainly related to ventricular fibrillation with arrhythmia. At present, there are few reports on the clinical and prognosis of ACS in China, and there is no guideline or consensus on the prevention and treatment of ACS patients. Known domestic research results show that the proportion of male, overweight / obese, smokers in young ACS patients is higher than that in the elderly group, while the proportion of patients with hypertension, diabetes and cerebrovascular diseases is less than that of the elderly group. The levels of TC, TG, LDL-C and UA and the proportion of low HDL-C in young ACS patients were higher than those in elderly patients; The diagnosis of STEMI was the highest in the young ACS group, while the diagnosis of unstable angina pectoris was the most common in the elderly ACS group. The clinical manifestations of ACS vary greatly. 3% ~ 5% of patients who exclude ACS only through myocardial markers, clinical blood transfusion and ECG still have myocardial infarction (MI). For the emergency department, early prediction of the risk of SCD in ACS patients and timely and accurate screening of high-risk patients are very important.

ELIGIBILITY:
Inclusion Criteria:

* The death event happens suddenly.
* Age ≥ 18 years
* The patient had obvious clinical symptoms 24 hours before treatment
* Life expectancy exceeds 3 days
* Proxy of patients signs the informed consent form
* Comply with ACS diagnostic indicators recommended by ACC / AHA guidelines in 2016

Exclusion Criteria:

* Death caused by accident, such as trauma, poisoning, etc.
* Death from accidental or intentional overdose
* Death from asphyxia
* Death is caused by chronic disease or terminal illness
* The patient died naturally
* Has participated in other clinical studies
* Immediate family members give up continuing treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sudden death
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence (or not of exosome-associated metabolites, microRNAs, and proteins | 2 years
  This outcome measure evaluates the presence (or not) of specific exosome-associated biomolecules, including metabolites (pyruvate, spermidine, glycine, glucose, L-phenylalanine), microRNAs (microRNA-208b-3p, microRNA-143-3p), and proteins (PSMB10, A1BG).

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China